CLINICAL TRIAL: NCT00935740
Title: Tissue Factor Expression in Stage C Heart Failure
Acronym: TFHF
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Mark A Munger, University of Utah
Other Study IDs: 5809-96; TFHF
Record Dates: First submitted 2009-06-18; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Heart Failure
Keywords: thromboembolic disease; thromboplastin; hypercoagulability; congestive heart failure
MeSH Terms: conditions — Heart Failure; Thromboembolism; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 50 ml of Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age-Matched Healthy Controls: Age-Matched Healthy Controls
- Heart Failure: Subjects with LVEF < 40%

SUMMARY:
Monocyte tissue factor (TF) was characterized in Class C heart failure (HF) vs. 25 age-matched volunteers. TF was 2.9 fold higher (p < 0.001) in HF patients vs. controls. HF patients showed increased clinical events (RR=1.29, p=0.04) when comparing procoagulant activity above/below median. HF is associated with increased TF expression.

DETAILED DESCRIPTION:
Monocyte tissue factor (TF) was characterized in Class C heart failure (HF) vs. 25 age-matched volunteers. TF was 2.9 fold higher (p < 0.001) in HF patients vs. controls. HF patients showed increased clinical events (RR=1.29, p=0.04) when comparing procoagulant activity above/below median. HF is associated with increased TF expression.

Previous studies suggest that markers of coagulation are elevated in heart failure (HF). Tissue factor (TF) plays the cardinal role in initiating the coagulation cascade. This study determines TF expression in HF and its association with disease progression.

Methods: Monocytes were obtained from 50 NYHA function class II-IV HF patients and 25 age-matched disease-free volunteers. TF protein, TF procoagulant activity, and tissue factor pathway inhibitor (TFPI) were determined.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure subjects with symptomatic heart failure (New York Heart Association [NYHA] functional class II to IV) due to either idiopathic dilated cardiomyopathy or ischemic cardiomyopathy and had a left ventricular ejection fraction < 0.35.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Heart failure
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 1996-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
This study determines TF expression in HF and its association with disease progression. | Hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Munger, Pharm.D., Principal Investigator — University of Utah